CLINICAL TRIAL: NCT04419727
Title: Molecular Analysis of Estrogen Receptors in Patients With Peripheral Artery Disease
Brief Title: Estrogen Receptors and Peripheral Artery Disease
Acronym: ESTROPAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Associate Professor of Vascular Surgery, University of Catanzaro
Other Study IDs: ER.ALL.2018.31
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Estrogen Deficiency; Peripheral Artery Disease
Keywords: Peripheral artery disease; Estrogens receptors; GPER
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: arterial reconstructive open surgery — Patients with peripheral artery disease (PAD) will undergo arterial reconstructive open surgery. Samples obtained from diseased arteries of lower limbs of patients undergoing arterial reconstructive open surgery will be collected and immediately preserved at -80°. Briefly, the arterial tissues will be excised, homogenized with a motor-driven homogenizer and total RNA will be isolated using Trizol reagent (Invitrogen, Milan Italy), according to the manufacturer's instructions. The expression of ER-alpha, ER-beta,and GPER will be quantified by real-time PCR using the Step One ™ sequence detection system (Applied Biosystems Inc. Milan, Italy), following the manufacturer's instruction

SUMMARY:
It is estimated that >200 million people have Peripheral artery disease (PAD) worldwide. PAD is related to increased morbidity or mortality in affected patients. More severe forms of PAD are surgically managed. Estrogen receptors (ERs) are strictly linked with vascular disease, and may be involved also in PAD onset and progression. This study will explore the expression of ERs, (ER-alpha, ER-beta,and a G protein-coupled of estrogen receptor -GPER-) in vessel wall of arteries of operated PAD patients, through the entire clinical spectrum of PAD.

DETAILED DESCRIPTION:
PAD is the atherosclerotic obstruction of the arteries of the lower extremities and it is widespread especially in highly developed countries. The most common complication of PAD is critical limb ischemia with rest pain and leg ulcers. To date the pathophysiology of PAD is linked to atherosclerosis but other pathways are also under evaluation. A recent study (Serra et al) investigated the presence of ER-alfa, ER-beta, and GPER in the wall of normal and varicose veins.

The aim of this observational study is to evaluate the expression and the role of estrogen receptors in patients with PAD, and undergoing surgical treatment with reconstructive arterial surgery. Therefore, we will collect tissue samples from diseased arteries that will be further analyzed for ER expression. We will then correlate the results with the clinical spectrum of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peripheral artery disease (PAD) eligible to receive arterial reconstructive open surgery.

Exclusion Criteria:

* malignancy
* estrogen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral artery disease (PAD) eligible to receive arterial reconstructive open surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-11-02 (Estimated)

PRIMARY OUTCOMES:
Expression of ER-alpha, ER-beta,and GPER | at month 6th
  The expression of ER-alpha, ER-beta,and GPER will be quantified by real-tome PCR using Step One ™ sequence detection system (Applied Biosystems Inc. Milan, Italy) following the manufacturer's instruction

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Serra, M.D., Ph.D., Principal Investigator — University Magna Graecia of Catanzaro
Locations (1):
- CIFL- Interuniversity Center of Phlebolymphology, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Criqui MH, Aboyans V. Epidemiology of peripheral artery disease. Circ Res. 2015 Apr 24;116(9):1509-26. doi: 10.1161/CIRCRESAHA.116.303849. PMID 25908725
- [Background] Serra R, Gallelli L, Perri P, De Francesco EM, Rigiracciolo DC, Mastroroberto P, Maggiolini M, de Franciscis S. Estrogen Receptors and Chronic Venous Disease. Eur J Vasc Endovasc Surg. 2016 Jul;52(1):114-8. doi: 10.1016/j.ejvs.2016.04.020. Epub 2016 May 21. PMID 27220899
- [Background] Barton M, Prossnitz ER. Emerging roles of GPER in diabetes and atherosclerosis. Trends Endocrinol Metab. 2015 Apr;26(4):185-92. doi: 10.1016/j.tem.2015.02.003. Epub 2015 Mar 9. PMID 25767029
- [Background] Boese AC, Kim SC, Yin KJ, Lee JP, Hamblin MH. Sex differences in vascular physiology and pathophysiology: estrogen and androgen signaling in health and disease. Am J Physiol Heart Circ Physiol. 2017 Sep 1;313(3):H524-H545. doi: 10.1152/ajpheart.00217.2016. Epub 2017 Jun 16. PMID 28626075
- [Background] Kublickiene K, Svedas E, Landgren BM, Crisby M, Nahar N, Nisell H, Poston L. Small artery endothelial dysfunction in postmenopausal women: in vitro function, morphology, and modification by estrogen and selective estrogen receptor modulators. J Clin Endocrinol Metab. 2005 Nov;90(11):6113-22. doi: 10.1210/jc.2005-0419. Epub 2005 Aug 30. PMID 16131583
- [Background] Kalicinska E, Wojtas K, Majda J, Zacharski M, Skiba J, Sliwowski J, Banasiak W, Ponikowski P, Jankowska EA. Expression of sex steroid receptors and aromatase in adipose tissue in different body regions in men with coronary artery disease with and without ischemic systolic heart failure. Aging Male. 2020 Jun;23(2):141-153. doi: 10.1080/13685538.2018.1494144. Epub 2018 Sep 7. PMID 30193537